CLINICAL TRIAL: NCT05233371
Title: Study of Parental Stress and Care Consumption Until 24 Months Corrected Age of Infants at a High Risk of Developmental Delay, After Discharge From Neonatal Intensive Care
Acronym: DeStreSs
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: KRUMM 2021-2
Record Dates: First submitted 2022-01-25; First posted 2022-02-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants at high risk of developmental delay
  Interventions: Other: Parenting Stress Index (PSI); Other: Collection of health care consumption; Other: Assessment of parent satisfaction

INTERVENTIONS:
Other: Parenting Stress Index (PSI) — collected by self-questionnaire during the follow-up carried out within the framework of the usual care (at 4, 9, 24 months of corrected age, +/- 18 months according to the neurodevelopmental evolution).
  Parental stress will be measured at each visit with the same parent (father or mother).
Other: Collection of health care consumption — Type and number of health professionals consulted between the different visits scheduled as part of the usual follow-up of the Dijon Bourgogne University Hospital,
  * Frequency and duration of rehabilitation sessions by type of health professionals,
  * Follow-up methods (institutional or private),
  Consumption of care will be evaluated by means of self-questionnaires given to parents during follow-up consultations as part of the usual care.
Other: Assessment of parent satisfaction — their level of information, their child's follow-up, and the support provided by the professionals.
  Satisfaction will be evaluated by means of a self-questionnaire (Likert scale) given to parents during follow-up consultations as part of their usual care.

SUMMARY:
Cerebral palsy (CP) is the leading cause of motor disability in children, affecting 125,000 people in France and with 1800 new cases per year. Prematurity remains a major risk factor, although children born at term represent 52% of children with cerebral palsy in France. Recent international and national (Haute Autorité de Santé, Troubles du neurodéveloppement - Repérage et orientation des enfants à risque, February 2020) recommendations emphasize the importance of continuous, early, and systematic management of infants at risk of cerebral palsy before 6 months of corrected age (CA), which is beneficial on the motor, cognitive, and social development of these children into preschool age. The principles of early identification and therapeutic intervention, which are at the core of multi-professional care, are becoming better known.

The priorities of this care are: the identification of high-risk infants, the continuity of follow-up from the neonatal period and after the return home in order to detect motor developmental disorders as early as possible, with a the global approach centered on the family. From the neonatal period, parents have traumatic experiences and are subjected to sources of stress. A framework of trust must be established during hospitalization, and preventive, multidisciplinary post-hospitalization follow-up is necessary. Informing families about the risks of motor developmental disorders that may affect their child and about the necessary follow-up in the first months is essential to obtain their adherence to an early course of action. This should take place even before parents have noticed abnormalities, and without waiting for a proven disability. However, it is necessary to support parents in these difficult situations by trying to reduce stress and to preserve the role of the parent.

Finally, the ESPaCe survey reveals several of the challenges faced by parents of children with CP: difficulty in finding trained therapists, low frequency of sessions, heterogeneity of rehabilitation techniques, and 75% of parents felt excluded from care and wish to be more involved. Fondation Motrice has therefore suggested developing recommendations for good clinical practice based on scientific evidence to address these difficulties.

In this context, the physiotherapists of the CHU Dijon Bourgogne have implemented the recommended early identification tools in the traditional perinatal follow-up pathway by collaborating with the neonatologists and rehabilitation physicians of the CHU Dijon Bourgogne. After the child goes home from the hospital, professionals can ensure continuity and adapt developmental support care by continuing to accompany the families. The follow-up pathway currently offered to these high-risk children includes a motor assessment at 4, 9 and 24 months of corrected age, with an additional consultation at 18 months of corrected age depending on the child's neurodevelopment. However, the psychological impact of this type of pathway on the parents, their satisfaction and their level of adherence to this care pathway are currently unknown.

Therefore, the objective of the DéStreSs study is to describe the level of parental stress and whether is varies over time, the consumption of care, parent satisfaction, and adherence to the follow-up program currently offered at the Dijon Bourgogne University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children hospitalized in the neonatal unit of the CHU Dijon and meeting at least one of the criteria below:
* Premature infants ≤ 31 weeks amenorrhea + 6 days
* And/or birthweight less than 1500 g,
* And/or children who presented with Intra-Ventricular Hemorrhage stages 3 or 4 according to the classification of Volpe et al. or Papile et al,
* And/or children who have had a cerebral vascular accident or anoxic-ischemic encephalopathy stage 2 or 3 according to the Sarnat classification,
* And/or children who have had a so-called serious condition during the neonatal period (i.e. cardiac or visceral surgery).

Exclusion Criteria:

* Parents who are minors,
* Parents under court protection,
* Parents of children with major orthopedic or traumatic disorders unrelated to neurodevelopmental risk,
* Parents unable to understand and respond to the questionnaires to be completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of children at high risk of developmental delay
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress Index (PSI) | throughout the visits until the child reaches 24 months of corrected age

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France